CLINICAL TRIAL: NCT05945082
Title: Presence of Fusobacterium Nucleatum at Colorectal Cancer Sites - Influencing Factors and Screening Possibilities
Brief Title: Fusobacterium Nucleatum at Colorectal Cancer Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malmö University (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Dnr 2016/469
Record Dates: First submitted 2023-07-03; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Periodontitis
MeSH Terms: conditions — Colorectal Neoplasms; Periodontitis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biopsy — biopsy of a colorectal cancer site

SUMMARY:
Recent studies suggest an association of periodontitis with an overall increased cancer risk but also with cancer development in specific anatomic regions, such as in the colon. The gut microbiome in general and specifically Fusobacterium nucleatum have been described to likely affect colorectal cancer (CRC) development. The present project intends to evaluate the possible contribution of the oral cavity as a reservoir for dissemination of F.nucleatum to the colon. Additionally, the gut microbiome and dietary intake will be assessed as possible factors influencing colonization of CRC sites with F. nucleatum and an association of F.nucleatum colonization in the colon with parameters in the saliva and serum will be tested. One-hundred-fifty patients diagnosed with CRC will be included; after cancer diagnosis and before starting cancer treatment a periodontal examination will be done and saliva and serum samples and at the time-point of tumor resection a biopsy of the CRC sites will be collected.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of colorectal cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of F.nucleatum in a colon cancer biopsy | At timepoint of biopsy
  dichotomous (present / absent)

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Plomp N, Bertl K, Lydrup ML, Sjoberg K, Harmsen HJM, Stavropoulos A. Does Fusobacterium in Colorectal Cancer Sites Originate From the Oral Cavity? A Pilot Study. Clin Exp Dent Res. 2024 Dec;10(6):e70016. doi: 10.1002/cre2.70016. PMID 39491831